CLINICAL TRIAL: NCT02826603
Title: A 52-week, Randomized, Double-blind Study of Secukinumab (300 mg) Compared to Ustekinumab in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Study of Secukinumab Compared to Ustekinumab in Subjects With Plaque Psoriasis
Acronym: CLARITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2326; 2015-002898-37 (EudraCT Number)
Record Dates: First submitted 2015-11-30; First posted 2016-07-11 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Plaque Psoriasis
Keywords: Plaque psoriasis; secukinumab; ustekinumab; ain457; ain457a
MeSH Terms: interventions — secukinumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): Secukinumab
  Interventions: Drug: Secukinumab
- Ustekinumab (Active Comparator): Ustekinumab
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Secukinumab — 300mg, s.c. at randomization, Weeks 1, 2 and 3 and thereafter 4-weekly till Week 48
  Arms: Secukinumab
Drug: Ustekinumab — Per approved label, 45 mg or 90 mg s.c. based on subject weight (at randomization visit) to be administered at randomization, Week 4, 16, 28 and 40. At other timepoints subjects will receive placebo injections.
  Arms: Ustekinumab

SUMMARY:
Demonstrate superiority of secukinumab over ustekinumab in treatment of moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give a written, signed and dated informed consent
* Chronic plaque-type psoriasis present for at least 6 months before randomization
* Moderate to severe plaque psoriasis as defined at randomization by:

  * PASI score of ≥12 and
  * Body Surface Area (BSA) affected by plaque-type psoriasis ≥10% and
  * IGA mod 2011 ≥3 (based on a scale of 0-4)
* Candidate for systemic therapy, defined as having psoriasis inadequately controlled by:

  * Topical treatment (including topical corticosteroids) and/or
  * Phototherapy and/or
  * Previous systemic therapy

Exclusion Criteria:

* Forms of psoriasis other than plaque psoriasis
* Drug-induced psoriasis
* Ongoing use of prohibited treatments
* Previous exposure to secukinumab or any other biologic drug directly targeting IL-17A or IL-17RA, or ustekinumab, or any therapies targeting IL-12 or IL-23
* Use of any other investigational drugs within 5 half-lives of the investigational treatment before study drug initiation
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1114 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (133):
- United States (106):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Glendale, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Fort Smith, Arkansas
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Rogers, Arkansas
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, California City, California
  - Novartis Investigative Site, Encinitas, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Irvine, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Santa Rosa, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Trumbull, Connecticut
  - Novartis Investigative Site, Aventura, Florida
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Cape Coral, Florida
  - Novartis Investigative Site, Coral Gables, Florida
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Orange Park, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Alpharetta, Georgia
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Newnan, Georgia
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, New Albany, Indiana
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Lake Charles, Louisiana
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Beverly, Massachusetts
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Brighton, Massachusetts
  - Novartis Investigative Site, Quincy, Massachusetts
  - Novartis Investigative Site, Fridley, Minnesota
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Saint Joseph, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, East Windsor, New Jersey
  - Novartis Investigative Site, Verona, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Forest Hills, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Rocky Mount, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dublin, Ohio
  - Novartis Investigative Site, Fairborn, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Oregon City, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Exton, Pennsylvania
  - Novartis Investigative Site, Jenkintown, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Plymouth Meeting, Pennsylvania
  - Novartis Investigative Site, Anderson, South Carolina
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Goodlettsville, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Murfreesboro, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Pflugerville, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Murray, Utah
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Everett, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Walla Walla, Washington
  - Novartis Investigative Site, Wenatchee, Washington
  - Novartis Investigative Site, Madison, Wisconsin
- Canada (4):
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Sainte-Hyacinthe, Quebec
- Czechia (2):
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (3):
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Kopavogur, Iceland
- Malaysia (2):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Johor Bahru
- Poland (5):
  - Novartis Investigative Site, Warsaw, Mazowian
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Warsaw
- Slovakia (2):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Bojnice
- South Korea (5):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Alpalhao M, Duarte J, Diogo R, Vandemeulebroecke M, Ortmann CE, Kasparek T, Filipe P. Lower Limbs are the Most Difficult-to-Treat Body Region of Patients with Psoriasis: Pooled Analysis of CLEAR and CLARITY Studies of Secukinumab Versus Ustekinumab by Body Region. BioDrugs. 2022 Nov;36(6):781-789. doi: 10.1007/s40259-022-00558-2. Epub 2022 Nov 5. PMID 36334236
- [Derived] Conrad C, Ortmann CE, Vandemeulebroecke M, Kasparek T, Reich K. Nail Involvement as a Predictor of Differential Treatment Effects of Secukinumab Versus Ustekinumab in Patients with Moderate to Severe Psoriasis. Dermatol Ther (Heidelb). 2022 Jan;12(1):233-241. doi: 10.1007/s13555-021-00654-1. Epub 2021 Dec 6. PMID 34870789
- [Derived] Bagel J, Blauvelt A, Nia J, Hashim P, Patekar M, de Vera A, Ahmad K, Paguet B, Xia S, Muscianisi E, Lebwohl M. Secukinumab maintains superiority over ustekinumab in clearing skin and improving quality of life in patients with moderate to severe plaque psoriasis: 52-week results from a double-blind phase 3b trial (CLARITY). J Eur Acad Dermatol Venereol. 2021 Jan;35(1):135-142. doi: 10.1111/jdv.16558. Epub 2020 Jun 8. PMID 32365251
- [Derived] Bagel J, Nia J, Hashim PW, Patekar M, de Vera A, Hugot S, Sheng K, Xia S, Gilloteau I, Muscianisi E, Blauvelt A, Lebwohl M. Secukinumab is Superior to Ustekinumab in Clearing Skin in Patients with Moderate to Severe Plaque Psoriasis (16-Week CLARITY Results). Dermatol Ther (Heidelb). 2018 Dec;8(4):571-579. doi: 10.1007/s13555-018-0265-y. Epub 2018 Oct 17. PMID 30334147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 1353 patients were screened of which 1102 patients completed the Screening phase; 251 patients were screen failures
Pre-assignment Details: The randomized set was defined as all patients who were randomized at the baseline visit. Unless otherwise specified, mis-randomized patients were excluded from the randomized set.
  Mis-randomized patients were those who were screen failures, but had been randomized by the Investigator before eligibility was assessed, but had not been treated
Groups:
- Secukinumab 300mg (2 x 150 mg): Secukinumab 300mg s.c. injection (2 150mg pre-fiilled syringes)
- Ustekinumab 2 x 45mg or 90mg: Ustekinumab s.c. 45 mg or 90 mg (depending on body weight) using 45mg pre-filled syringes (1 or 2 syringes)
Period: Overall Study
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Started | 550 | 552
Completed | 489 | 488
Not Completed | 61 | 64
Not completed — Adverse Event | 17 | 9
Not completed — Lack of Efficacy | 4 | 9
Not completed — Lost to Follow-up | 13 | 12
Not completed — Noncompliance with treatment | 0 | 2
Not completed — Physician Decision | 1 | 7
Not completed — Pregnancy | 1 | 2
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 20 | 19
Not completed — Death | 2 | 0
Not completed — New therapy for study indication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg | Total
Number analyzed (Participants) | 550 | 552 | 1102
Age, Continuous [Mean (Standard Deviation); unit: years] — average age of participants
  years | 45.4 (14.09) | 45.3 (14.16) | 45.4 (14.12)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 488 | 494 | 982
  >=65 years and <75 years | 60 | 48 | 108
  >=75 years | 2 | 10 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 176 | 370
  Male | 356 | 376 | 732
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 416 | 410 | 826
  Black | 21 | 24 | 45
  Asian | 60 | 57 | 117
  Native American | 34 | 41 | 75
  Pacific Islander | 1 | 5 | 6
  Unknown | 4 | 2 | 6
  Other | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response at Week 12
Description: Number of participants who achieved ≥ 90% reduction in PASI compared to baseline.
  Logistic regression analysis of PASI 90 response at Week 12
  PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, upper limbs, trunk, lower limbs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of body region(head: 0.1, upper limbs: 0.2, trunk: 0.3, lower limbs: 0.4).
Time Frame: Week 12
Population: The Full analysis set (FAS) is all patients from the randomized set assigned to study treatment. Following the intent-to-treat principle, patients were analyzed according to the treatment assigned at randomization. If the actual randomization stratum was different to the assigned stratum in IRT, the actual stratum was used in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Number analyzed (Participants) | 550 | 552
Participants | 366 | 265
Statistical Analysis 1: Comparison: Secukinumab 300mg (2 x 150 mg) vs Ustekinumab 2 x 45mg or 90mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.72 to 2.84]

2. Primary Outcome: Participants With IGA Mod 2011 0 or 1 at Week 12
Description: Investigator's Global Assessment uses a scale (IGA mod 2011) that rates disease from a score of 0 (clear skin) to 4 (severe disease)
Time Frame: Week 12
Population: The full analysis set (FAS) population was used for this analysis. The FAS included all participants to whom treatment was assigned. Only participants from the FAS, who had values at a given week, were included in the analysis for that week.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Number analyzed (Participants) | 550 | 552
Participants | 397 | 306
Statistical Analysis 1: Comparison: Secukinumab 300mg (2 x 150 mg) vs Ustekinumab 2 x 45mg or 90mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.10, 95% CI 2-sided [1.63 to 2.72]

3. Secondary Outcome: Participants Who Achieved Psoriasis Area and Severity Index (PASI) 75 Response at Week 12
Description: Number of participants who achieved ≥ 75% reduction in PASI at Week 12 compared to baseline.
Time Frame: Week 12
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Number analyzed (Participants) | 550 | 552
Participants | 484 | 409
Statistical Analysis 1: Comparison: Secukinumab 300mg (2 x 150 mg) vs Ustekinumab 2 x 45mg or 90mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.89 to 3.62]

4. Secondary Outcome: Participants Who Achieved Psoriasis Area and Severity Index (PASI) 75 Response at Week 4
Description: Number of participants who achieved ≥ 75% reduction in PASI at Week 4 compared to baseline.
Time Frame: Week 4
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Number analyzed (Participants) | 550 | 552
Participants | 221 | 90
Statistical Analysis 1: Comparison: Secukinumab 300mg (2 x 150 mg) vs Ustekinumab 2 x 45mg or 90mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.53, 95% CI 2-sided [2.65 to 4.71]

5. Secondary Outcome: Participants Who Achieved Psoriasis Area and Severity Index (PASI) 100 Response at Week 16
Description: Number of participants who achieved 100% reduction in PASI at Week 16 compared to baseline.
Time Frame: Week 16
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Number analyzed (Participants) | 550 | 552
Participants | 250 | 147
Statistical Analysis 1: Comparison: Secukinumab 300mg (2 x 150 mg) vs Ustekinumab 2 x 45mg or 90mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.80 to 3.01]

6. Secondary Outcome: Participants With IGA Mod 2011 0 or 1 at 16 Weeks
Description: as for outcome 2
Time Frame: Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Number analyzed (Participants) | 550 | 552
Participants | 432 | 326
Statistical Analysis 1: Comparison: Secukinumab 300mg (2 x 150 mg) vs Ustekinumab 2 x 45mg or 90mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.96 to 3.37]

7. Secondary Outcome: Participants Who Achieved Psoriasis Area and Severity Index (PASI) 100 Response at Week 12
Description: Number of participants who achieved 100% reduction in PASI at Week 12 compared to baseline.
Time Frame: Week 12
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Number analyzed (Participants) | 550 | 552
Participants | 210 | 111
Statistical Analysis 1: Comparison: Secukinumab 300mg (2 x 150 mg) vs Ustekinumab 2 x 45mg or 90mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.50, 95% CI 2-sided [1.89 to 3.31]

8. Secondary Outcome: Participants Who Achieved Psoriasis Area and Severity Index (PASI) 75 Response at Week 16
Description: Number of participants who achieved ≥ 75% reduction in PASI at Week 16 compared to baseline.
Time Frame: Week 16
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Number analyzed (Participants) | 550 | 552
Participants | 506 | 441
Statistical Analysis 1: Comparison: Secukinumab 300mg (2 x 150 mg) vs Ustekinumab 2 x 45mg or 90mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.86, 95% CI 2-sided [1.96 to 4.17]

9. Secondary Outcome: Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response at Week 16
Description: Number of participants who achieved ≥ 90% reduction in PASI at Week 16 compared to baseline.
Time Frame: Week 16
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Number analyzed (Participants) | 550 | 552
Participants | 423 | 299
Statistical Analysis 1: Comparison: Secukinumab 300mg (2 x 150 mg) vs Ustekinumab 2 x 45mg or 90mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.85, 95% CI 2-sided [2.19 to 3.71]

10. Secondary Outcome: Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response at Week 52
Description: Number of participants who achieved ≥ 90% reduction in PASI at Week 52 compared to baseline.
Time Frame: Week 52
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300mg (2 x 150 mg) | Ustekinumab 2 x 45mg or 90mg
Number analyzed (Participants) | 550 | 552
Participants | 402 | 330
Statistical Analysis 1: Comparison: Secukinumab 300mg (2 x 150 mg) vs Ustekinumab 2 x 45mg or 90mg; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.41 to 2.41]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for approximately 52 months. All cause mortality (deaths) was collected from First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV) up to a maximum of 52 weeks
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 52 weeks
Groups:
- AIN457 300 mg: Secukinumab 300mg s.c. injection in 2 150mg pre-fiilled syringes
- UST 45/90 mg: Ustekinumab s.c. 45mg or 90 mg (depending on body weight) (using 45mg pre-filled syringes)
- All Patients: All Patients from both arms
Arm/Group | AIN457 300 mg | UST 45/90 mg | All Patients
All-Cause Mortality (participants affected / at risk) | 2/550 | 0/552 | 2/1102
Serious Adverse Events (participants affected / at risk) | 29/550 | 21/552 | 50/1102
Other Adverse Events (participants affected / at risk) | 216/550 | 229/552 | 445/1102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg (N=550) | UST 45/90 mg (N=552) | All Patients (N=1102)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 1
Colitis erosive (Gastrointestinal disorders) | 1 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2 | 3
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1
Dengue fever (Infections and infestations) | 2 | 0 | 2
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Skin candida (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Device inappropriate shock delivery (Product Issues) | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Renal infarct (Renal and urinary disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg (N=550) | UST 45/90 mg (N=552) | All Patients (N=1102)
Diarrhoea (Gastrointestinal disorders) | 26 | 24 | 50
Nausea (Gastrointestinal disorders) | 6 | 13 | 19
Bronchitis (Infections and infestations) | 8 | 18 | 26
Conjunctivitis (Infections and infestations) | 12 | 6 | 18
Nasopharyngitis (Infections and infestations) | 55 | 54 | 109
Sinusitis (Infections and infestations) | 25 | 18 | 43
Upper respiratory tract infection (Infections and infestations) | 49 | 61 | 110
Urinary tract infection (Infections and infestations) | 13 | 9 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 14 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 20 | 34
Headache (Nervous system disorders) | 26 | 25 | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 16 | 33
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 17 | 31
Dermatitis contact (Skin and subcutaneous tissue disorders) | 12 | 8 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 18 | 30
Hypertension (Vascular disorders) | 17 | 22 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT02826603/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT02826603/SAP_001.pdf